CLINICAL TRIAL: NCT01880229
Title: Phase II and Phase IIB STTR: Portable Device for Telecare Monitoring of Elderly People
Brief Title: Physical Activity Monitoring in Frailty and Falling
Status: Completed | Type: Observational
Sponsor: BioSensics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: 12-0659-01; 2R42AG032748 (NIH)
Record Dates: First submitted 2013-06-14; First posted 2013-06-18 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Fraility; Risk of Falling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- non-frail: Categorized as non-frail based on Fried's five phenotypic criteria (Fried L.P., et al. Frailty in Older Adults: Evidence for a Phenotype. Journal of Gerontology: 2001, Vol. 56A, No. 3, M146-M156)
- pre-frail: Categorized as pre-frail based on Fried's five phenotypic criteria (Fried L.P., et al. Frailty in Older Adults: Evidence for a Phenotype. Journal of Gerontology: 2001, Vol. 56A, No. 3, M146-M156)
- frial: Categorized as frail based on Fried's five phenotypic criteria (Fried L.P., et al. Frailty in Older Adults: Evidence for a Phenotype. Journal of Gerontology: 2001, Vol. 56A, No. 3, M146-M156)

SUMMARY:
BioSensics has developed a Physical Activity Monitoring System (PAMSys) that consists of a single wearable motion sensor that is worn on the torso. The objectives of this observational study are the following: 1) to test the efficacy of PAMSys for objectively assessing a persons risk of falling based on activity data measured during activities of daily living and 2) to test the efficacy of PAMSys for identifying precise early physical activity or functioning indicators of frailty in those who are pre-frail or frail as compared to non-frail controls.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling ambulatory men or women ages 65 and above

Exclusion Criteria:

* Mental Status Mini Exam score < 23
* Those who are unwilling or unable to comprehend informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Pima County Arizona elders aged 65+ will be recruited from the Arizona Center on Aging affiliated geriatrics clinics.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-08; Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Average sit-to-stand transition time over 48-hour monitoring period | Averaged over days 1 and 2
  Eligible subjects will receive a PAMSys motion sensors and necessary instructions for proper use. They will then wear the motion sensor continuously for 48 hours. PAMSys will record the duration of each sit-to-stand transition during this 48 hour monitoring period. The primary outcome measure is the average of these durations.

SECONDARY OUTCOMES:
Average stand-to-sit transition time during 48 hours of continuous monitoring | Averaged over days 1 and 2
  Eligible subjects will receive a PAMSys motion sensors and necessary instructions for proper use. They will then wear the motion sensor continuously for 48 hours. PAMSys will record the duration of each stand-to-sit transition during this 48 hour monitoring period. The primary outcome measure is the average of these durations.

OTHER OUTCOMES:
Fraility as categorized based on Fried's five phenotypic criteria | First evaluation (day 1)
  Fried L.P., et al. Frailty in Older Adults: Evidence for a Phenotype. Journal of Gerontology: 2001, Vol. 56A, No. 3, M146-M156
Fraility as categorized based on Fried's five phenotypic criteria | 6 months
  Fried L.P., et al. Frailty in Older Adults: Evidence for a Phenotype. Journal of Gerontology: 2001, Vol. 56A, No. 3, M146-M156

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Gwin, PhD, Principal Investigator — BioSensics; Bijan Najafi, PhD, Principal Investigator — University of Arizona; Jane Mohler, PhD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona Center on Aging, Tucson, Arizona
  - Baylor College of Medicine Interdisciplinary Consortium on Advance Motion Performance, Houston, Texas

REFERENCES:
- [Derived] Pradeep Kumar D, Najafi B, Laksari K, Toosizadeh N. Sensor-Based Assessment of Variability in Daily Physical Activity and Frailty. Gerontology. 2023;69(9):1147-1154. doi: 10.1159/000530900. Epub 2023 May 10. PMID 37231977
- [Derived] Pradeep Kumar D, Wendel C, Mohler J, Laksari K, Toosizadeh N. Between-day repeatability of sensor-based in-home gait assessment among older adults: assessing the effect of frailty. Aging Clin Exp Res. 2021 Jun;33(6):1529-1537. doi: 10.1007/s40520-020-01686-x. Epub 2020 Sep 15. PMID 32930988
- [Derived] Pradeep Kumar D, Toosizadeh N, Mohler J, Ehsani H, Mannier C, Laksari K. Sensor-based characterization of daily walking: a new paradigm in pre-frailty/frailty assessment. BMC Geriatr. 2020 May 6;20(1):164. doi: 10.1186/s12877-020-01572-1. PMID 32375700
- [Derived] Parvaneh S, Mohler J, Toosizadeh N, Grewal GS, Najafi B. Postural Transitions during Activities of Daily Living Could Identify Frailty Status: Application of Wearable Technology to Identify Frailty during Unsupervised Condition. Gerontology. 2017;63(5):479-487. doi: 10.1159/000460292. Epub 2017 Mar 11. PMID 28285311